CLINICAL TRIAL: NCT05930249
Title: Effect of a fNIRS-based Personalized Multi-domain Intervention on Cognitive in Elderly Population With High Risk of Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FNIRS
Record Dates: First submitted 2023-06-06; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Impairment; Stroke; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Stroke; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard health counseling (No Intervention)
- Personalized multidomain intervention (Experimental)
  Interventions: Behavioral: Personalized multidomain intervention

INTERVENTIONS:
Behavioral: Personalized multidomain intervention — 1. Patients will complete personalized cognitive training based on baseline fNIRS on APP (20-30 mins/day, 3-4 days/week, 6 months).
  2. Shared decision-making on risk factor of stroke between doctors and patients
  3. Social support by grouping patients online to ensure close interaction with other patients in the same arm
  Arms: Personalized multidomain intervention

SUMMARY:
This functional near-infrared spectroscopy-based personalized multidomain intervention study aims to prevent cognitive impairment and reduce dementia and cerebrovascular events in 45-74 years old persons with high risk of stroke in China. The primary outcome is 6-months change in global cognitive score measured by a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network protocol. The investigators hypothesize that the intervention based on functional near-infrared spectroscopy will prevent cognitive decline by the initial 6-months intervention. The long-term primary outcome is the development of dementia and cerebrovascular events during a total of 2 years' follow-up. The investigators hypothesize that the functional near-infrared spectroscopy-based personalized intervention may reduce the 2-year risk of dementia and cerebrovascular events, mainly through the improvement in vascular risk factors control, social activity, and cognitive training activities.

DETAILED DESCRIPTION:
Patients with ≥ 3 stroke risk factors (including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke), or with transient ischemic attack, are regarded as patients with high risk of stroke. Studies have indicated that these stroke risk factors might be associated with an increased risk of cerebral small vessel disease (CSVD) progress, glymphatic dysfunction, cognitive decline, dementia, and cerebrovascular events. However, prevention in these patients is largely unknown and the management of these patients is a very troublesome issue. Management on those patients mainly focused on improving lifestyle. Recently, cognitive training has emerged, with change from strategy-oriented paper-and-pencil and instructional training methods to computer-aided cognitive training that is difficulty adaptive and focuses on ability improvement. Studies have shown that the functional state of the brain is more sensitive and specific than the behavioral performance, so it provides a theoretical basis for personalized intervention. Functional near-infrared spectroscopy imaging converts signal values into oxygenated hemoglobin, deoxyhemoglobin, and changes in overall hemoglobin concentration according to Beer-Lambert's law to reflect brain activity levels, which is more convenient than EEG and functional magnetic resonance in collecting task-state signal. By pre-analyzing the correlation between the activation level of each brain region and cognition, the brain area related to cognitive function under each task can be preliminarily obtained, and the patient can be further judged whether the patient needs to be trained for the task according to the activity level of the brain region to achieve the purpose of personalization. The investigators hypothesize that the intervention based on functional near-infrared spectroscopy imaging will reduce cognitive impairment, CSVD progress, and reduce dementia and cerebrovascular events incidence in the study group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-74 years
* high risk of stroke (with≥3 of 8 stroke risk factors, including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke, or with transient ischemic attack)

Exclusion Criteria:

* previously diagnosed dementia
* previously diagnosed stroke (both cerebral infarction and hemorrhage)
* suspected dementia after clinical assessment by study physician at screening visit
* Mini-mental State Examination [MMSE] score<20
* disorders affecting safe engagement in the intervention (e.g., malignant disease, major depression, symptomatic cardiovascular disease, revascularization within 1 year previously)
* severe loss of vision, hearing, or communicative ability
* disorders preventing cooperation as judged by the study physician
* coincident participation in another intervention trial
* any MRI contraindications

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network protocol | 6 months
  Primary Outcome

SECONDARY OUTCOMES:
Cognitive domain change assessed with NINDS-CSN protocol, including working memory, executive function, language, visual motor speed, visual spatial function, memory and recognition | 6 months
  short-term secondary outcome
Cognitive domain change assessed with NINDS-CSN protocol, including working memory, executive function, language, visual motor speed, visual spatial function, memory and recognition | 2 year
  long-term secondary outcome
Cognitive function change assessed by Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive function change assessed by Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 year
  long-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 year
  long-term secondary outcome
Signal change of resting-state functional near-infrared spectroscopy | 6 months
  short-term secondary outcome
Signal change of resting-state functional near-infrared spectroscopy | 2 year
  long-term secondary outcome
Activation changes of task functional near-infrared spectroscopy | 6 months
  short-term secondary outcome
Activation changes of task functional near-infrared spectroscopy | 2 year
  long-term secondary outcome
Changes in image markers (WMHs, lacunes, microbleeds, perivascular spaces, brain atrophy, micro-infarcts) of CSVD assessed on MRI | 6 months
  short-term secondary outcome
Changes in image markers (WMHs, lacunes, microbleeds, perivascular spaces, brain atrophy, micro-infarcts) of CSVD assessed on MRI | 2 year
  long-term secondary outcome
Changes in functional network-related characteristics assessed by fMRI, including intra- and inter-network connectivity, graph theory, and dynamic functional connectivity | 6 months
  short-term secondary outcome
Changes in functional network-related characteristics assessed by fMRI, including intra- and inter-network connectivity, graph theory, and dynamic functional connectivity | 2 year
  long-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 6 months
  short-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 2 year
  long-term secondary outcome
Changes in metabolite composition to measure the change of metabolite profiles in participants' faecal samples and serum samples | 6 months
  short-term secondary outcome; metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Changes in metabolite composition to measure the change of metabolite profiles in participants' faecal samples and serum samples | 2 year
  long-term secondary outcome; metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)

CONTACTS AND LOCATIONS:
Locations (1):
- Min Lou, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided